CLINICAL TRIAL: NCT00027287
Title: Preliminary Assessment of Laser and Medical Treatment of Diabetic Macular Edema
Brief Title: Laser and Medical Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020063; 02-EI-0063
Record Dates: First submitted 2001-11-29; First posted 2001-11-30 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-12

CONDITIONS: Diabetes Mellitus; Macular Edema
Keywords: Type I Diabetes; Type 2 Diabetes; Diode Laser Photocoagulation; Vitamin E; Elevated Low-Density Lipoprotein (LDL-C) Cholesterol; Diabetic Retinopathy; Macular Edema; Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Retinopathy | interventions — Vitamin E

INTERVENTIONS:
Drug: Vitamin E

SUMMARY:
This study will compare the side effects of two laser treatments for diabetic macular edema, a common condition in patients with diabetes. In macular edema, blood vessels in the retina-a thin layer of tissue that lines the back of the eye-become leaky and the retina swells. The macula-the center part of the retina that is responsible for fine vision-may also swell and cause vision loss. Traditional laser treatment (argon blue or green or yellow) for macular swelling, or edema, causes scarring that can expand and possibly lead to more loss of vision. Studies with a different type of laser (diode) have shown no adverse effects to the retina, but long-term effects of this treatment are not known. The results of this study on side effects of the treatments will be used to design a larger study of effectiveness. This study will also examine whether vitamin E can reduce the damage caused by laser treatment. Patients with diabetic eye disease who take vitamin E have increased blood flow through the vessels of the retina, as well as improved kidney function. Patients with elevated cholesterol levels will be invited to participate in a cholesterol reduction part of the study to compare normal-pace cholesterol reduction with accelerated reduction.

Patients 18 years of age and older with type 1 or type 2 diabetes and macular edema may be eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history - to review past medical conditions and treatments.
* Physical examination - to measure vital signs (pulse, blood pressure, temperature, breathing rate) and examine the head and neck, heart, lungs, abdomen, arms and legs.
* Eye examination - to assess visual acuity (eye chart test) and examine pupils, lens, retina, and eye movements. The pupils will be dilated with drops for this examination.
* Blood tests - to measure cholesterol and vitamin E blood levels, blood clotting time, hemoglobin A1C (a measure of diabetes control), and to evaluate liver and kidney function.
* Photography - to help evaluate the status of the retina and changes that may occur in the future. Special photographs of the inside of the eye are taken using a camera that flashes a bright light into the eye. From 2 to 20 pictures may be taken, depending on the eye condition.
* Fluorescein angiography - to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.

Participants will be randomly assigned to receive one of the two laser treatments. They will also be randomly assigned to take 1600 IU of vitamin E or placebo (an inactive, look-alike pill) daily. For the laser treatment, eye drops are put in the eye to numb the surface and a contact lens is placed on the eye during the laser beam application. Several visits may be required for additional laser treatments. The maximum number of treatments depends on how well the treatment is working.

On their first visit, patients will be given vitamin C. After taking the vitamin for 1 month, they will return to the clinic for the first laser treatment. They will followed 1, 3, 6, 9, and 12 months after the first treatment, and then every 6 months until either 1) the patient returns for a 3-year visit; 2) the last enrolled patient returns for the 1-year visit, or the patient requests to leave the study. During these visits, several of the exams described above will be repeated to evaluate the response to treatment and check for side effects of the vitamin E.

DETAILED DESCRIPTION:
This randomized pilot study is an important first step in planning a large multi-center clinical trial to evaluate medical and laser approaches that could improve the visual outcome for patients with diabetic retinopathy. This study will provide preliminary safety data on these therapies as well as allow for assessment of the performance of ocular outcomes and study design for use in subsequent trials. If there are no safety concerns, the results of this pilot will be helpful in the design of a large multicenter clinical trial by providing data on estimates of expected treatment effects. A larger trial will proceed regardless of whether or not this study identifies statistically significant main effects.

Using a partial factorial design, this study will compare (1) diode (micropulse) laser photocoagulation to mild ETDRS style focal photocoagulation and, (2) treatment with Vitamin E, a COX-2 inhibitor (celecoxib), or placebo prior to and following laser photocoagulation. The primary safety outcome is a visual acuity drop of 15 letters or more from baseline one year following initial laser treatment. The primary efficacy outcome will be reduction of the retinal thickening defined as an improvement by at least two steps (on standard fundus photos) combined with a 50% reduction in the area of fluorescein leakage one year after the initial laser compared to baseline. A secondary outcome will be the change in macular height as measured (OCT). These outcomes will be assessed for potential use in future trials. Concerns regarding safety and efficacy follow:

Safety

Is the risk of visual loss in patients with clinically significant diabetic macular edema potentially different across treatment groups?

Preliminary Assessment of Potential Outcomes

Is there evidence that any treatment combinations could be effective in reducing retinal thickening?

Is there evidence that Vitamin E may affect the ability of either photocoagulation method to reduce retinal thickening, or vice versa?

Is there evidence that celecoxib may inhibit retinal thickening?

What are the estimated treatment effects on vision?

Is the number of laser treatments required to achieve a reduction in retinal thickening similar across treatment groups?

A tertiary objective of this study will be to examine the effects of dramatically reducing low-density lipoproteins cholesterol in patients with diabetic macular edema and elevated serum lipids. Change vision and retinal thickness will be compared across three groups; (1) patients without elevated serum lipids at baseline, (2) patients with elevated lipids at baseline and receive standard of care treatment, and (3) patients with elevated lipids at baseline and are aggressively treated pharmacologically.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with type 1 or 2 diabetes.

Patients with clinically significant macular edema in at least one eye.

Best corrected visual acuity 20/400 or better as measured on an ETDRS chart in the eye with clinically significant macular edema; this eye will be considered the study eye. If both eyes have clinically significant macular edema and best corrected visual acuity greater than or equal to 20/400, the right eye will be considered the study eye.

May have had proliferative diabetic retinopathy but scatter photocoagulation must be performed more than six months ago.

Ocular media sufficiently clear to allow for quality fundus photography.

If Aphakic or pseudophakic, lens removal must have occurred at least 6 months prior to enrollment.

Clinical diagnosis of diabetes based on any one of the criteria (determined by medical physician):

Documented history of plasma glucose value greater than 210 mg/dl on 3 different occasions.

Fasting blood sugar greater than 150 mg/dl on 3 different occasions.

Documented history of ketoacidosis.

Insulin dependency.

Documented history of abnormal glucose tolerance test.

Patient's medical status must include a likelihood of survival for 5

years.

Hemoglobin A1C 12 percent or less.

Willingness to accept randomization for diet or drug therapy for lowering of elevated lipid levels.

Understand and sign the informed consent.

Patients over 18 years of age since the population of interest is primarily older than 18.

A negative urine pregnancy test for women of childbearing potential.

EXCLUSION CRITERIA:

Retinopathy that requires scatter photocoagulation immediately.

Ocular disease other than diabetic retinopathy that may confound the outcome of the study (e.g. age-related macular degeneration, drug toxicity, uveitis, etc.).

Had previous focal laser photocoagulation for diabetic macular edema.

Poor survival due to other systemic diseases (separate from diabetes)

Poor glycemic control with hemoglobin A1C greater than 12 percent.

Past or current liver disease, which precludes the use of the lipid-lowering drugs.

Vitamin E supplementation over and above the amount in a multivitamin (30 IU/day) one month prior to entry into the study.

History of hypersensitivity to fluorescein.

History of intra-cranial bleeds.

Evidence of other ocular diseases that may confound the assessment of treatment of diabetic macular edema.

Prior or current macular detachment in the affected eye(s).

Concurrent celebrex or any other COX-2 inhibitor within 7 days prior to baseline.

Concurrent coumadin therapy or known bleeding diathesis.

Concurrent treatment with a new investigational drug.

Concurrent lithium therapy

Malabsorption syndrome.

Concurrent administration of anti-cholesterol resin medications (e.g. cholestyramine)

Concurrent administration of the anti-obesity drug orlistat (Xenical).

Concurrent administration of other NSAIDs.

Allergy to sulphonomides, NSAIDs, or exhibit the aspirin triad.

Pregnant or lactating women.

Chronic requirement for any ocular medication for other diseases such as glacoma.

Current history of malignancy (except patients having a basal cell carcinoma that was treated successfully, or other malignancy operated on and in remission for 5 years prior to inclusion in the trial).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2001-11; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] The effect of intensive diabetes treatment on the progression of diabetic retinopathy in insulin-dependent diabetes mellitus. The Diabetes Control and Complications Trial. Arch Ophthalmol. 1995 Jan;113(1):36-51. doi: 10.1001/archopht.1995.01100010038019. PMID 7826293
- [Background] Grattagliano I, Vendemiale G, Boscia F, Micelli-Ferrari T, Cardia L, Altomare E. Oxidative retinal products and ocular damages in diabetic patients. Free Radic Biol Med. 1998 Aug;25(3):369-72. doi: 10.1016/s0891-5849(98)00059-8. PMID 9680184